CLINICAL TRIAL: NCT06999122
Title: Multi-Center, Prospective, Consecutive, Paired Diagnosis, Diagnostic Performance Study of the EMVision Emu™ Brain Scanner in the Detection of Intracranial Hemorrhage in Suspected Stroke Patients
Brief Title: Diagnostic Performance Study of the EMVision Emu™ Brain Scanner in the Detection of Intracranial Hemorrhage in Suspected Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: EMVision Medical Devices Ltd (Network)
Responsible Party: Sponsor
Other Study IDs: EMV-CIP-03
Record Dates: First submitted 2025-05-13; First posted 2025-05-31 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Hemorrhagic Stroke
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Intracranial Haemorrhage Group A
  Interventions: Diagnostic Test: Brain Scan
- Other Group B: Group B includes all patients enrolled in the study ultimately diagnosed with a condition other than intracranial haemorrhage, including ischaemic stroke, transient ischaemic attack, or any of a variety of stroke mimicking conditions.
  Interventions: Diagnostic Test: Brain Scan

INTERVENTIONS:
Diagnostic Test: Brain Scan — The EMVision emu™ Brain Scanner is a device system which scans the human brain using radiofrequency techniques. The emu™ headset is placed on the head of a patient, enabling ultra-high frequency radio wave (also commonly referred to as microwave) signal propagation into the patient's head.
  The radio-waves reflect from and transmit through the tissue boundaries and are detected by the receiver antennae within the headset. The transceivers operate at very low-level signals in accordance with national and international safety thresholds. The scattered signals carry information on the scanned tissues.

SUMMARY:
The purpose of this research is to evaluate a new investigational device for the diagnosis of stroke, the EMVision emu™ Brain Scanner. Stroke is the result of a blood clot stopping the normal flow of blood in the brain (ischaemic stroke) or a breakage in a blood vessel causing bleeding in the brain (haemorrhagic stroke). Stroke is a medical emergency and must be quickly diagnosed and treated. Computed tomography (CT) or magnetic resonance imaging (MRI) scans are commonly used to diagnose stroke, but they are not always readily available.

EMVision has developed the emu™ Brain Scanner, a helmet-like device which scans the head using ultra-high frequency radio signals. It is portable and easy to use, making it more accessible than CT or MRI machines. Easier access to the EMVision emu™ Brain Scanner may reduce the time taken to diagnose stroke, leading to faster treatment and better health outcomes. It is the purpose of this study in the first instance to determine the accuracy of the EMVision emu™ Brain Scanner in the detection of haemorrhagic stroke.

DETAILED DESCRIPTION:
This clinical investigation is a paired diagnosis, diagnostic performance study intended to quantify the accuracy of the emu™ Brain Scanner's diagnostic output in comparison to current gold-standard practices including multi-modal neuroimaging by CT and/or MRI.

Any adult with neurological deficit suspected to be stroke presenting to the investigational site's emergency department shall be considered as potentially eligible for the study. Potential participant's eligibility for the study is determined via screening evaluation which includes a review of available demographic and medical history information against the study's inclusion and exclusion criteria, as well as a head size assessment using provided gauges to confirm that their head would fit within the emu™ Brain Scanner. If the screening evaluation finds that the participant is eligible for the study then the investigator proceeds with the informed consent process. This activity occurs in parallel with the investigational site's standard practices for stroke patient management, ensuring no delay in these patients' care.

Regardless of study participation, participants will receive the complete standard of care diagnostic workflow in accordance with applicable national and international guidelines, as well as practices established at the investigational site. The standard of care diagnostic workflow is centered around acute baseline multi-modal CT imaging (and in some instances MRI). Directly following or before this imaging, and without delaying subsequent treatment, a scan is completed with the emu™ Brain Scanner to allow timely coordination between the investigational emu™ Brain Scan result and the reference standard CT/MRI imaging. If the attending physician perceives any potential risk of delaying treatment of the patient then that patient is strictly exclude from the study, entirely at the attending physician's discretion.

A central adjudicating ground truth diagnosis panel is formed of experts in the area of stroke diagnosis and reviews all diagnostic information gathered by the investigational site as per the site's standard of care diagnostic workflow. The ground truth diagnosis panel is blinded to the output from the emu™ Brain Scanner and defines the 'ground truth' or 'reference standard' diagnosis for each patient to ensure accuracy and consistency. Integral to the ground truth diagnosis panel's consideration is the assessment by the core imaging lab, who similarly review all imaging provided by the investigational sites to ensure consistent input to the ground truth expert panel.

The result of the emu™ Brain Scan is compared to the ground truth diagnosis by a biostatistician to determine the accuracy of the emu™ Brain Scanner's diagnostic output (in terms of sensitivity and specificity) with the first output evaluated being intracranial haemorrhage detection in suspected stroke patients. The biostatistician then performs all statistical analyses against the study objectives in accordance with the Statistical Analysis Plan.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥22 years of age
2. Presenting to hospital with acute neurological deficit suspected to be stroke and within 12 hours of symptom onset
3. The use of the EMVision emu™ Brain Scanner will not delay the treatment of the patient
4. CT or MRI brain imaging following clinical evaluation in Emergency Department per standard of care
5. Head size deemed suitable for scanning with the EMVision emu™ Brain Scanner -

Exclusion Criteria:

1. Has received treatment for current (suspected) stroke event prior to initial CT/MRI scan OR EMVision emu™ Brain Scanner scan (such as thrombolysis)
2. Contraindication to neuroimaging, such as a contrast allergy or other condition that prohibits CT, MRI and/or angiography
3. Presence of any implanted electro-stimulating devices in the head and neck
4. Presence of any metallic implants in the cranial vault or surrounding bones/tissue (Note that metallic objects distant from the scan area, such as dental implants, nasal piercing etc., are acceptable)
5. Presence of an intracranial pressure monitor or any other similar sensor that may compromise the placement of the investigational device
6. Inability to wear the investigational device (skin lesions on scalp, obvious recent blunt or penetrating injury to head, previous intracranial surgeries, neck injury etc.)
7. Unable to lie still for the duration of the scan
8. Pregnant or breastfeeding
9. Any other condition or symptoms preventing the participant from entering the study, according to the investigator´s judgment -

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 subjects across two study arms
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Demonstrate haemorrhage detection sensitivity >80% and specificity >80% | <30 minutes from acute baseline CT/MRI

SECONDARY OUTCOMES:
Demonstrate the time to complete an emu™ Brain Scan is <15 minutes | <30 minutes from acute baseline CT/MRI
Evaluate safety of the device | <30 minutes from acute baseline CT/MRI
Evaluate usability of the device | <30 minutes from acute baseline CT/MRI
Evaluate device deficiencies | <30 minutes from acute baseline CT/MRI

CONTACTS AND LOCATIONS:
Overall Officials: Reade De Leacy, MBBS(Hons) FRANZCR, Principal Investigator — Associate Professor of Neurosurgery and Radiology Director of Neurointerventional Spine Site Director Cerebrovascular Services Mount Sinai Queens Co-director Neuroendovascular Surgery Fellowship Department of Neurosurgery Mount Sinai Health System; Angela Dos Santos, PhD, Principal Investigator — Melbourne Health
Locations (4):
- United States (2):
  - Mayo Jacksonville, Jacksonville, Florida
  - UTHealth, Houston, Texas
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Melbourne Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT06999122/ICF_000.pdf